CLINICAL TRIAL: NCT01069562
Title: Comparison of Isoflurane Anaesthesia by Closed Loop Controlled Administration Versus Manually Controlled Administration Using Bispectral Index in Open Heart Surgery
Brief Title: Closed Loop Isoflurane Administration With Bispectral Index in Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Prof G. D. Puri, Post Graduate Institute of Medical Education and Research
Organization: PIMERIndia (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: closed loop isoflurane
Record Dates: First submitted 2010-02-01; First posted 2010-02-17 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2010-07

CONDITIONS: Open Heart Surgery
Keywords: closed loop control of anesthesia; isoflurane; open heart surgery

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- MANUAL (Active Comparator): In the manual group isoflurane was administered using Tech 7 vapouriser. The dial setting was controlled by the anesthesiologist to achieve and maintain a BIS of 50 during anesthesia.
  Interventions: Other: Conventional control
- IAADS group (Experimental): In this group, liquid isoflurane was injected into the circuit using a syringe pump controlled by the IAADS system.The IAADS system has the algorithm to regulate the rate of infusion of isoflurane such that BIS is achieved and maintained at 50 during anesthesia.
  Interventions: Other: Closed loop control

INTERVENTIONS:
Other: Conventional control — The isoflurane administration to deliver anesthesia will be done conventionally through a Tec 7 vaporiser to maintain the bispectral index at 50.
  Other Names: MANUAL CONTROL
  Arms: MANUAL
Other: Closed loop control — The isoflurane administration to maintain anesthesia will be by infusion to the anesthesia circuit using syringe pump (injection technique). The rate of delivery of isoflurane will be regulated by computer that uses a control algorithm.
  Other Names: AUTOMATED CONTROL
  Arms: IAADS group

SUMMARY:
With the advancement in microprocessor technology and better understanding of pharmacodynamics and pharmacokinetics of anaesthetic agents, computer facilitated closed loop control of anaesthesia using propofol has been shown to be accurate with better performance than manual control. Literature on computer controlled administration of inhalational anaesthetics is few, as it requires the computer to control the dial setting on the vapouriser. The investigators intend to compare the computer controlled closed loop administration of isoflurane by infusing it into the anaesthetic circuit with conventional vaporiser control in elective open heart surgery.

40 patients (ASA (American Society of Anesthesiology) class II-IV; 18- 65 years) undergoing elective cardiac surgery requiring cardiopulmonary bypass (CPB) will be randomly divided into manual or closed loop groups. Propofol will be used for induction of anaesthesia in both groups followed by isoflurane for maintenance. In the manual group, isoflurane will be administered through the Tech 7 vapouriser during pre and post CPB periods to target bispectral index (BIS) of 50. In closed loop group, isoflurane will be administered using infusion of liquid isoflurane into expiratory limb of the closed circuit. This rate of infusion though a conventional syringe pump will be controlled by algorithm termed 'Improvised Anaesthetic Agent Delivery System' (IAADS) to maintain BIS of 50. Patients in both groups will receive 500ml of 100 % oxygen as fresh gas flow. The % of time bispectral index (BIS) is within the 10 of set target BIS of 50 will be the primary outcome measure. The secondary outcome measures will be median performance error (MDPE)(2), median absolute performance error (MDAPE)(2), wobble(2), divergence(2), amount of isoflurane used and hemodynamic parameters will be secondary outcome measures.

DETAILED DESCRIPTION:
The basic components in a closed loop anesthesia delivery system are: (1) a system under control- patient; (2) a controlled variable that measures depth of anesthesia, (3) a set point for this variable specified by the user, (4) an actuator which comprises an algorithm to translate a measured value of the controlled variable to a particular action or the actuator to steer the controlled variable closer to the target variable.

In the proposed study, the controlled variable will be BIS. The control actuator is a patented (2158/DEL/2007) pharmacodynamic- pharmacokinetic model based adaptive infusion system termed "Improved Anesthetic Agent Delivery System (IAADS"). An IBM compatible with PENTIUM 2 or higher processor personal computer (2 GHz) is used to implement the control algorithm, provide a user interface and control communication through serial ports (RS 232) with the infusion system (Pilot- C, Frasenius, France) and a Datex vital sign monitor. We will use Avance ventilator (Datex Ohmeda, software version 5.0) with carbon di oxide absorber and ascending bellows to provide constant volume ventilation. The amount of acceptable leak in the circuit will be reduced to ≤ 150 ml min-1 determined during ventilation of a test lung. Low fresh gas flows will be used during the study. Isoflurane will injected into the expiratory limb of circle system via 20 ml Plastipak (polyethylene BD) syringe with a 100 cm long polyethylene tubing (Vygon, India) using a Pilot C Infusion pump (Fresenius vial SA, France). The stated volumetric accuracy of the infusion pump is ±2 %.

After obtaining written informed consent, patients will be randomly allocated (by closed envelope technique using computer generated random numbers) to one of the two groups- manual and automatic. The investigator will be present during the procedure for data collection purpose only and will not be involved in the conduct of anaesthesia. All patients will receive 5- 10mg oral diazepam as per institutional protocol the night before and on the morning of surgery as pre-medication. After shifting the patient to the operation table, patients will be started on normal saline 100 ml/hr (1-2 ml/kg/hr). Routine physiological monitoring will be commenced (pulse oximetry, electrocardiography, non-invasive blood pressure monitoring). BIS (Bispectral index)will be obtained by disposable sensors (Aspect medical system Inc. MA USA) attached to the forehead of the patient. Patients will receive 0.15 mg/kg of morphine sulphate before induction in aliquots of 3-5mg, during which indwelling arterial cannula, central venous line and pulmonary artery catheters (if deemed to be necessary) will be inserted.

Before induction, patients shall receive fentanyl 3μg/kg over three minutes. In automatic mode, IAADS automatically will calculate and titrate the initial and subsequent propofol infusion rate according to the weight of the patient, risk status and target BIS value, which will be set at 50 for all cases with a range of 40-60. In manual group, the propofol infusion rate will be determined by the attending anaesthesiologist according to the weight of the patient, and the target BIS of 50, with the aim to maintain BIS within 40- 60. After loss of consciousness (LOC), patients will receive 0.1mg/kg vecuronium bromide and will be intubated after 4 minutes.

The circle system will be closed after ascertaining the correct position of the endotracheal tube. In the control group, isoflurane infusion will be started into the expiratory limb of the circle at predetermined rates. The isoflurane concentration in the circuit will be built gradually over a period of 10 minutes to attain a specified BIS value. During isoflurane anaesthesia, patients will be ventilated with 100% oxygen. Fresh gas flows will be started at 500ml/min, and the ventilation will be set so as to maintain an end tidal CO2 concentration of 30-35 mmHg. If the fresh gas flows are inadequate as determined by incomplete filling of bellows, the flows will be increased gradually by 100 ml/min till a maximum of 1000 ml/min. If still there is a leak, the study will be abandoned and patient ventilated with higher flows. Thus, patients will be maintained on isoflurane injected into the expiratory limb of the circuit. Analgesia will be maintained with fentanyl 1μg/kg/hr infusion with further boluses of 1μg/kg before skin incision, sternotomy and commencement of cardiopulmonary bypass (CPB). Muscular relaxation will be maintained with a continuous infusion of vecuronium bromide 50μg/kg/hr. After 30 minutes of induction, an arterial sample will be drawn to have baseline values for blood gases, activated clotting time (ACT), and blood glucose. Patients will receive a bolus of 3 mg/kg heparin to raise the ACT above 480s. In cases of lower values, further boluses of heparin will be infused as per bull and colleagues dose response curve for heparin.

In the manual group, after the confirmation of the placement of endotracheal tube, the circle system will be closed and fresh gas flows will be started at 1000ml/min. Inhalational anaesthetics will be delivered by Fluotech 7 vapouriser (Datex ohmeda) for isoflurane. The initial dial setting will be started at 3% and after 5 minutes, flows will be reduced to 500 ml/min and isoflurane concentration will be titrated by the anaesthesiologist to maintain BIS of 50. The dial setting will be increased or decreased to maintain BIS of 50 and the number of times the vapouriser dial setting is changed will be noted. Rest of the protocol will be similar to the computer control group described above.

After the initiation of CPB, arterial blood gases, ACT and blood glucose will be determined every half an hour. An arterial partial pressure of O2 of 300-400 mmHg, ACT >480s and blood glucose <180mg/dl will be maintained throughout the bypass period. After successful completion of cardiopulmonary bypass, heparin will be antagonised with protamine sulphate.

During episodes when the mean arterial pressure exceeds 25% of the baseline or heart rate exceeds 100 beats/ min or 25% of the baseline, analgesia will be supplemented with fentanyl 1μg/kg. In case of persistent hypertension or tachycardia with BIS < 50, nitroglycerine infusion will be started and titrated to control blood pressure; Esmolol (upto 0.5mg/kg IV) will be administered to control the heart rate (HR). Similarly, in case of fall in mean arterial pressure to less than 25% of the baseline in the presence of normovolemia, initially phenylephrine will be used in boluses of 0.5μg/kg. For persistent hypotension after a cumulative Phenylephrine dose of 2μg/kg, dopamine infusion will be started and titrated to maintain MAP within 25% of the baseline. Likewise, in case of decrease in HR to <45beats/min., atropine sulphate (10μg/kg IV boluses) will be administered after excluding other treatable causes.

During CPB, patients will be shifted to propofol infusion, as the equipment for delivering fresh gases during CPB requires large fresh gas flows and circle system is not possible presently. MAP will be maintained between 50- 80 mmHg and any deviation from theses limits shall be treated with Phenylephrine boluses or sodium nitroprusside infusion. Propofol will be administered as per IAADS in computer control group and manually in the manual group to maintain BIS of 50.

Five minutes after the end of CPB, patients will be shifted back to isoflurane. In the computer control group, the concentration in the circuit for the set BIS will be achieved over 10 minutes. In the manual control group, the dial setting will be started at 3% and titrated according to the BIS. Fresh gas flows will be maintained at the same rate before the initiation of CPB.

At the end of skin closure, isoflurane, fentanyl and vecuronium will be stopped and the study protocol terminated. Patient will be shifted to propofol infusion for post operative sedation and will be shifted to post anaesthesia care unit without antagonizing muscle relaxants for elective mechanical ventilation. Patients will be extubated on meeting standard criteria for extubation. All patients will be continuously monitored for hemodynamic stability and maintenance of blood gases upto 24 hrs postoperatively. Patients will be subjected to a structured interview as modified from Brice and colleagues and described by Nordstrom for conscious awareness; on discharge from post anesthesia care unit, the day after surgery and approximately a week later.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology physical status 2- 4
* elective open heart surgery under general anaesthesia
* requiring Cardio Pulmonary Bypass (CPB)

Exclusion Criteria:

* body weight ±30% of the ideal body weight
* neurological disorder
* use of any psychoactive medication
* severe stenotic valve lesions
* severe pulmonary artery hypertension
* Tetrology of Fallot repair and other cyanotic heart diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Puri GD, MBBS MD PhD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Sethu Madhavan, MBBS, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Preethy J Mathew, MBBS, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Post graduate institute of medical education and research, Chandigarh, India

REFERENCES:
- [Background] Locher S, Stadler KS, Boehlen T, Bouillon T, Leibundgut D, Schumacher PM, Wymann R, Zbinden AM. A new closed-loop control system for isoflurane using bispectral index outperforms manual control. Anesthesiology. 2004 Sep;101(3):591-602. doi: 10.1097/00000542-200409000-00007. PMID 15329583
- [Background] Varvel JR, Donoho DL, Shafer SL. Measuring the predictive performance of computer-controlled infusion pumps. J Pharmacokinet Biopharm. 1992 Feb;20(1):63-94. doi: 10.1007/BF01143186. PMID 1588504
- [Background] Agarwal J, Puri GD, Mathew PJ. Comparison of closed loop vs. manual administration of propofol using the Bispectral index in cardiac surgery. Acta Anaesthesiol Scand. 2009 Mar;53(3):390-7. doi: 10.1111/j.1399-6576.2008.01884.x. PMID 19243324
- [Background] Puri GD, Kumar B, Aveek J. Closed-loop anaesthesia delivery system (CLADS) using bispectral index: a performance assessment study. Anaesth Intensive Care. 2007 Jun;35(3):357-62. doi: 10.1177/0310057X0703500306. PMID 17591128
- [Derived] Madhavan JS, Puri GD, Mathew PJ. Closed-loop isoflurane administration with bispectral index in open heart surgery: randomized controlled trial with manual control. Acta Anaesthesiol Taiwan. 2011 Dec;49(4):130-5. doi: 10.1016/j.aat.2011.11.007. Epub 2011 Dec 22. PMID 22221684

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment of participants started on 10th January 2009 and ended on 24th June 2010. All patients recruited were admitted for elective cardiac surgery in the Cardio Thoracic Surgery ward in Post Graduate Institute of Medical Education and Research, Chandigarh, India.
Pre-assignment Details: All the patients who were enrolled were randomized to the two study arms.
Groups:
- Manual: The manual group in which isoflurane will be administered using Tech 7 vapouriser. The dial setting will be controlled by the anesthesiologist.
- IAADS Group: In this group, liquid isoflurane will be injected into the circuit using a syringe pump controlled by the IAADS system.
Period: Overall Study
Arm/Group | Manual | IAADS Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Manual | IAADS Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 46.4 (15.2) | 46.4 (14.1) | 46.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 14 | 16 | 30
Region of Enrollment [Number; unit: participants]
  India | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Time Bispectral Index Remains Within 10 of Target BIS of 50
Description: The duration of time depth of anesthesia was maintained in the recommended range (as measured by BIS) during the period isoflurane (general anesthetic) was administered to the study population. This value expressed as percentage is the primary outcome. BIS is an objective measure of depth of anesthesia derived from statistical(bispectral) analysis of electroencephalographic waves. BIS ranges from 0 to 100. It decreases monotonically from 100 in the awake state to lower values with sedation and anesthesia.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
percentage of time | 75.9 (11.2) | 84.6 (7.2)

2. Secondary Outcome: Median Performance Error (MDPE)
Description: The difference between the observed and target of measure of depth of anesthesia (BIS) expressed as percentage of target BIS is calculated as performance error every 30 seconds. This value may be either '+' or '_' indicating whether the observed measure is above the target (overshoot-+) or below the target (undershoot-_). The median value of all performance errors during isoflurane anesthesia is median performance error and is a measure of bias of the system. This outcome is expressed as the mean of Median Performance Errors per participant.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: percentage deviation of BIS from target
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
percentage deviation of BIS from target | 7.5 (7.3) | 4.8 (4.9)

3. Secondary Outcome: Median Absolute Performance Error (MDAPE)
Description: The median of the absolute values of performance errors (without considering the direction of error) is median absolute performance error. This outcome measures the magnitude of error or inaccuracy of the system studied. A lower value indicates a more precise system.This outcome is expressed as the mean of Median Absolute Performance Errors per participant.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: percentage deviation of absolute BIS
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
percentage deviation of absolute BIS | 13.2 (3.7) | 11.0 (2.7)

4. Secondary Outcome: Wobble
Description: Wobble measures the intra-individual variability in performance error.The median of the difference between individual performance errors throughout anesthesia and the median performance error for each participant is the wobble of that participant. The mean value per participant is indicated in the outcome measure.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: percentage of BIS
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
percentage of BIS | 9.3 (3.5) | 8.7 (1.7)

5. Secondary Outcome: Percentage of Time Heart Rate Remained Within 25% of Pre-op Baseline
Description: The duration of time heart rate remained within 25% of the pre-operative baseline value during the period isoflurane (general anesthetic) was administered to the study population. This value is expressed as a percentage. This outcome is expressed as the mean of percentage of time per participant.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
percentage of time | 77.3 (17.6) | 86.1 (10.4)

6. Secondary Outcome: Percentage of Time Mean Arterial Pressure Remained Within 25% of Pre-op Baseline
Description: The duration of time mean arterial pressure remained within 25% of the pre-operative baseline value during the period isoflurane (general anesthetic) was administered to the study population. This value is expressed as percentage. This outcome is expressed as the mean of percentage of time per participant
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
percentage of time | 76.0 (17.2) | 80.4 (9.8)

7. Secondary Outcome: Intra-operative Awareness
Description: The number of patients who were able to recall the intra-operative events when assessed postoperatively. This was assessed by a structured protocol
Time Frame: 3 days (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Number; unit: participants
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
participants | 0 | 0

8. Secondary Outcome: Fentanyl Used
Description: The total amount of fentanyl that was used during the procedure.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: µg/kg
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
µg/kg | 10.1 (1.4) | 10.1 (1.2)

9. Secondary Outcome: Intra Operative Adrenaline Used
Description: The amount of adrenaline used during the procedure
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: µg/kg
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
µg/kg | 2.6 (0.4) | 2.7 (0.3)

10. Secondary Outcome: INTRA OPERATIVE PHENYLEPHRINE USED
Description: The amount of phenylephrine used during the procedure.
Time Frame: 8 hours (approximately)
Population: All the patients who were randomized completed the study protocol and were included for analysis
Measure: Mean (Standard Deviation); unit: .µg/kg
Arm/Group | Manual | IAADS Group
Number analyzed (Participants) | 20 | 20
.µg/kg | 5.2 (1.4) | 4.5 (1.5)

ADVERSE EVENTS:
Arm/Group | Manual | IAADS Group
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 3/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Manual (N=20) | IAADS Group (N=20)
High inotropic requirement intra-op (Cardiac disorders) | 3 (3) | 2 (2) — The number of patients who required a dose ≥ 0.1 µg/kg/min of adrenaline infusion for any duration of time or addition of a second inotropic agent during cardiac surgery.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes